CLINICAL TRIAL: NCT02465983
Title: Pilot Study of Autologous T-cells Redirected to Mesothelin and CD19 With a Chimeric Antigen Receptor in Patients With Metastatic Pancreatic Cancer
Brief Title: Pilot Study of Autologous T-cells in Patients With Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy and funding to continue investigation
Sponsor: University of Pennsylvania (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 19214, 821275; UPCC 19214 (Other: University of Pennsylvania Cancer Center); UCSF CC144520 (Other: University of California San Francisco Cancer Center)
Record Dates: First submitted 2015-05-28; First posted 2015-06-09 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; CAR / CART; T cells; Immunotherapy; Gene therapy; Redirected T cells; Autologous T cells
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CART-meso-19 T cells (Experimental): A single dose of CART-meso-19 T cells (combination therapy with CART-meso and CART19 cells) will be administered intravenously as two separate infusions. The dose is 1-3x107/m2 (Cohort 1) or 1-3x108/m2 (Cohort 2) CART positive cells. The infusion will be scheduled to occur 3 (±1) days after a single dose of 1.5 grams/m2 of cyclophosphamide, which will be administered according to standard procedures in the outpatient setting.
  Interventions: Biological: CART-meso-19 T cells; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: CART-meso-19 T cells — A single dose of CART-meso-19 cells (combination therapy with CART-meso and CART19 cells) will be administered intravenously as two separate infusions. The dose is 1-3x107/m2 (Cohort 1) or 1-3x108/m2 (Cohort 2) CART positive cells. The infusion will be scheduled to occur 3 (±1) days after a single dose of 1.5 grams/m2 of cyclophosphamide, which will be administered according to standard procedures in the outpatient setting. Patients will receive CART cell treatment on an outpatient basis.
Drug: Cyclophosphamide — A single dose of chemotherapy to be administered prior to dosing of the CART-meso-19 cells

SUMMARY:
This is a study in which pancreatic cancer patients receive a combination therapy with CART-meso cells and CART19 cells administered at 3 days after one dose of cyclophosphamide. CART-meso cells are patients' own T cells that were modified in the laboratory to express a receptor specific to the mesothelin protein. CART19 cells are patients' own T cells that were modified in the laboratory to express a receptor specific to a protein called CD19. The CD19 protein is expressed on white blood B cells. CART19 cells are expected to attack the B cells and impede the antibody response against CART-meso cells. The investigators hypothesize that this combination therapy may prolong the duration of CART-meso cells in the body. Additionally, one dose of cyclophosphamide may enhance engraftment and persistence of CART cells.

DETAILED DESCRIPTION:
Immunotherapy is a novel and promising approach for the treatment of solid tumors; immunotherapy with chimeric antigen receptor (CAR) T cells (CART cells) in particular has the potential advantage of targeted therapies that can invoke a rapid tumor response, and the advantage of long-lived responses that are the hallmark of engagement of the adaptive immune system such as memory T cells.

This is a single arm, open-label, phase I study to determine the safety and feasibility of combination CART-meso cells (autologous T cells lentivirally transduced to express anti-mesothelin scFv fused to TCRζ and 4-1BB costimulatory domains) and CART19 cells (autologous T cells lentivirally transduced to express a humanized anti-CD19 scFv fused to TCRζ and 4-1BB costimulatory domains) in patients with pancreatic cancer following lymphodepletion with cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Unresectable or metastatic pancreatic cancer
* Persistent cancer after at least one prior standard of care chemotherapy for advanced stage disease
* 18 years of age and older
* ECOG performance status of 0 or 1
* Life expectancy greater than 3 months
* Satisfactory organ and bone marrow function
* Meets blood coagulation parameters
* Male and Female subjects of reproductive potential agree to use approved contraceptive methods

Exclusion Criteria:

* Participation in a therapeutic investigational study within 4 weeks prior to the screening visit
* Anticipated need for systemic chemotherapy within 2 weeks before apheresis and infusion
* Active invasive cancer other than pancreatic cancer
* HIV, HCV, or HBV infections
* Active autoimmune disease requiring immunosuppressive therapy within 4 weeks prior to screening visit, with exception of thyroid replacement
* Ongoing or active infection
* Planned concurrent treatment with systemic high dose corticosteroids
* Patients requiring supplemental oxygen therapy
* Prior therapy with gene modified cells
* Previous experimental therapy with SS1 moiety, murine or chimeric antibodies
* History of allergy to murine proteins
* History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40)
* Clinically significant pericardial effusion, CHF, or cardiovascular condition that would preclude assessment of mesothelin induced pericarditis or that may worsen as a result of toxicities expected for this study
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-05; Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Safety of IV administration of CART-meso-19 with cyclophosphamide as lymphodepleting chemotherapy in patients with pancreatic cancer using the NCI CTCAE v4.03 criteria | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Plesa, Study Director — University of Pennsylvania; Andrew Ko, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States